CLINICAL TRIAL: NCT02121522
Title: A Single Arm Open Label Study to Evaluate the Pharmacodynamics and Safety of a 4 wk Treatment With BI 144807 in Patients With Newly Diagnosed Wet Age Related Macular Degeneration (wAMD)
Brief Title: A 4 Week Study With BI 144807 in Patients >= 50 Years With Wet Age Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1313.20; 2013-004567-30 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Wet Macular Degeneration
MeSH Terms: conditions — Wet Macular Degeneration

ARMS (1):
- BI 144807 (Experimental): twice daily
  Interventions: Drug: BI 144807

INTERVENTIONS:
Drug: BI 144807 — twice daily

SUMMARY:
The present trial will use an open label design to investigate the effect of BI 144807 on central 1-mm retinal thickness and presence of neovascular leakage in newly diagnosed wAMD patients. A further objective is to collect data on adverse events, vital signs, ECG and clinical laboratory parameters of BI 144807 in the same patient group.

ELIGIBILITY:
Inclusion criteria:

Newly diagnosed men and women with unilateral subfoveal choroideal neovascularization secondary to age-related macular degeneration

Exclusion criteria:

Additional eye disease that could compromizse best corrected visual acuity, such as uncontrolled glaucoma

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- 1313.20.43001 Boehringer Ingelheim Investigational Site, Vienna, Austria
- Germany (6):
  - 1313.20.49004 Boehringer Ingelheim Investigational Site, Bonn
  - 1313.20.49002 Boehringer Ingelheim Investigational Site, Leipzig
  - 1313.20.49001 Boehringer Ingelheim Investigational Site, Lübeck
  - 1313.20.49005 Boehringer Ingelheim Investigational Site, Münster
  - 1313.20.49003 Boehringer Ingelheim Investigational Site, Tübingen
  - 1313.20.49006 Boehringer Ingelheim Investigational Site, Ulm
- Hungary (3):
  - 1313.20.36002 Boehringer Ingelheim Investigational Site, Budapest
  - 1313.20.36003 Boehringer Ingelheim Investigational Site, Budapest
  - 1313.20.36001 Boehringer Ingelheim Investigational Site, Debrecen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a open-label, single-arm, 4-week proof-of-concept study.
Groups:
- BI 144807: Subjects were orally administered with 400 mg film coated tables twice daily (two tablets of 200 mg twice daily)
Period: Overall Study
Arm/Group | BI 144807
Started | 14
Completed | 13
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients who were dispensed study medication and were documented to have taken at least one dose of study drug.
Arm/Group | BI 144807
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in CRT as Measured by SD-OCT on Day 29
Description: Change from baseline in central 1-mm retinal thickness (CRT) as measured by spectral domain optical coherence tomography (SD-OCT) on day 29.
Time Frame: Baseline (day 1) and day 29
Population: Treated set (WOCF). Missing values are imputed by the worst observation carried forward (WOCF) measurement (including baseline).
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | BI 144807
Number analyzed (Participants) | 14
μm | 44.0 (151.5)

2. Secondary Outcome: Change From Baseline in Neovascular Leakage Area as Assessed by FA on Day 29
Description: Change from baseline in neovascular leakage area as assessed by Fluorescein angiography (FA) on day 29. Baseline is defined as the last value collected before the first trial drug intake. Data collected after start of wet age-related macular degeneration (wAMD) therapy are set to missing.
Time Frame: Baseline and day 29
Population: Treated set (OC). Observed Case (OC): This method analysed only available data that were observed while patients were on treatment, ie., missing data were not imputed.
Measure: Mean (Standard Deviation); unit: mm²
Arm/Group | BI 144807
Number analyzed (Participants) | 10
mm² | -0.7 (1.4)

ADVERSE EVENTS:
Time Frame: From first drug administration until 5 days after last drug administration, up to 5 weeks.
Arm/Group | BI 144807
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 144807 (N=14)
Retinal haemorrhage (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 144807 (N=14)
Retinal haemorrhage (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Body temperature increased (Investigations) | 1
Headache (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The trial was ended earlier as per protocol as the preliminary data showed that the likelihood to meet the trial's primary efficacy endpoint would have been low even if the patient recruitment had been continued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.